CLINICAL TRIAL: NCT01987297
Title: Combined Retinoic Acid,Arsenic Trioxide and Chemotherapy for Newly-diagnosed Acute Promyelocytic Leukemia: Chinese National Multi-center Randomized Study
Brief Title: Combined Retinoic Acid,Arsenic Trioxide and Chemo for Newly-diagnosed APL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Tang-Du Hospital (Other); Peking University People's Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); First Hospital of China Medical University (Other); Southwest Hospital, China (Other); West China Hospital (Other); Ningbo No. 1 Hospital (Other); Qilu Hospital of Shandong University (Other); Shandong Provincial Hospital (Other Government); Union hospital of Fujian Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Guangdong Provincial People's Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Jiong HU, Department of Hematology, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL2012
Record Dates: First submitted 2012-12-06; First posted 2013-11-19 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: acute promyelocytic leukemia; ATRA; arsenic
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Tretinoin; Arsenic Trioxide; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATRA+Arsenic (Experimental): All low- and intermediate-risk patients receive retinoic acid and arsenic trioxide based consolidation. High-risk patients receive ATRA+Arsenic+Anthracycline consolidation.
  Interventions: Drug: ATRA+Arsenic
- ATRA+chemo (Active Comparator): All low-risk and intermediate-risk patients receive retinoic acid and chemotherapy with idarubicin or daunorubicin as consolidation. High-risk patients receive ATRA+anthracycline and cytarabine as consolidation.
  Interventions: Drug: ATRA+Chemo

INTERVENTIONS:
Drug: ATRA+Arsenic — ATRA: 25mg/m2 daily；Induction: D1 to CR; Consolidation: D1-14 each course; Maintenance: D1-14 each course.
  Arsenic: 0.16mg/kg daily. Induction: D1 to CR; Consolidation: low/intermediate-risk patients 28 days each course; high-risk: 14 days each course; Maintenance: 14 days on and off each course.
  Idarubicin 8mg/m2 or Daunorubicin 45mg/m2 daily. Induction: 3-4 days in high-risk patients or intermediated-risk patients with leukocytosis developed during induction therapy. Consolidation: 3 days in high-risk patients in first 2 courses.
  MTX: 15mg/m2 qw Maintenance: qw x 4 in each course for high-risk patients.
  Other Names: retinoic acid + arsenic trioxide
  Arms: ATRA+Arsenic
Drug: ATRA+Chemo — ATRA: 25mg/m2 daily；Induction: D1 to CR; Consolidation: D1-14 each course; Maintenance: D1-14 each course.
  Arsenic: 0.16mg/kg daily. Induction: D1 to CR; Maintenance: 14 days on and off each course.
  Idarubicin 8mg/m2 or Daunorubicin 45mg/m2 daily. Induction: 3-4 days in high-risk patients or intermediated-risk patients with leukocytosis developed during induction therapy. Consolidation: 3 days in all patients in 2 courses.
  Cytarabine: 150mg/m2 or 1g/m2. Consolidation: 150mg/m2 daily x 7 days in high risk patients in first 2 courses; 1g/m2 q12 x 6 doses in third course.
  MTX: 15mg/m2 qw Maintenance: qw x4 in each course for high-risk patients.
  Other Names: retinoic acid + idarubicin or daunorubicin +/- Cytarabine
  Arms: ATRA+chemo

SUMMARY:
In this prospective randomized study for patients with newly diagnosed acute promyelocytic leukemia, patients will be randomized (1:1) into two groups which receive retinoic acid and arsenic trioxide based treatment versus retinoic acid and chemotherapy based regimen.

DETAILED DESCRIPTION:
The study is carried out based on Sanz risk stratification of newly-diagnosed APL patients into low-, intermediate- and high-risk groups, and all of them will receive ATRA and ATO as induction therapy (ATRA 25 mg/m2 per day orally + ATO 0.16mg/kg intravenously daily). Anthracycline is added to both high-risk groups or intermediate-risk group with hyperleukocytosis developed during induction therapy but not in low-risk groups.

After achieving CR, patients enter into consolidation therapy. Low-risk patients receive either 2 courses of ATRA plus ATO (Experimental group) or 2 courses of ATRA plus anthracycline chemotherapy (Control group). Intermediate-risk patients receive either 3 courses of ATRA plus ATO (Experimental group) or 2 courses of ATRA plus anthracycline chemotherapy (Control group). Patients of high-risk disease receive 2 courses of ATRA plus ATO and anthracycline and 1 course of ATRA plus ATO treatment (Experimental group) or 2 courses of ATRA plus anthracycline and cytarabine and 1 course of ATRA plus mid-dose cytarabine (Control group).

After consolidation therapy, patients with molecular complete remission (mCR) enter into maintenance therapy. Low- and intermediate-risk patients receive 3 cycles of ATRA and ATO sequential treatment, while those of high-risk receive 5 cycles of ATRA, ATO and methotrexate (MTX) treatment.

For low- and intermediate-risk patients who fail to achieve mCR after consolidation therapy, 3 courses of consolidation therapy of high-risk group will be given with cross-over (i.e. patients in Experimental group received the therapy of Control group, and patients in Control group received the therapy of Experimental group). If patients still fail to achieve mCR, together with high-risk group who fail to achieve mCR after consolidation therapy will be withdrawn from the study and proceed to salvage treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed patients with acute promyelocytic leukemia via cytogenetics and molecular assay
* Age: 18-65
* Hepatic/renal function: Bil≤35μmol/L，AST/ALT less than 2Xnormal range, Cr 150μmol/L
* Normal cardial function
* ECOG：0-4
* Informed consent

Exclusion Criteria:

* QTC interval >450ms
* Pregnant or breast feeding patients
* Patients with drug addiction or mental illness
* Patients documented of CNS infiltration at diagnosis
* Patients with severe heart disease (acute myocardial infarction or heart failure)
* Patients with concurrent active malignancy, tuberculosis or HIV infection
* Patients with contraindication or allergy to anthracyclines or other agent in the protocol
* Patients enrolled in other clinical trials
* Patients not apply to the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 3 year
  DFS is defined for patients having achieve CR as time to relapse either in bone marrow or extra medullary site, or fail to achieve molecular remission, or death of all causes.

SECONDARY OUTCOMES:
Complete remission (CR) rate | after induction therapy
  Blast and promyelocytic leukemia less than 5% in bone marrow
Molecular CR (mCR) | after consolidation therapy
  mCR is defined the absence of detectable PML-RARα transcripts by nested RT-PCR or RQ-PCR in two successive bone marrow samples
Early death (ED) rate | 30 days
  Early death is referred to death within 30 days from the entry into the treatment.
Overall survival (OS) | 3 years
  OS is defined for patients entering the study as time to death of all causes.
Cumulated incidence of relapse (CIR) | 3 years
  CIR is defined for patients having achieved CR as time to any relapse or persistence of PCR positivity after consolidation therapy

OTHER OUTCOMES:
Hematological or non hematological toxicitytoxicitie | 3 years
  Assessed according to the Common Terminology Criteria for Adverse Events Version 4.0 (National Cancer Institute)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-min Li, M.D, Principal Investigator — Department of Hematology, Rui Jin Hospital, Shanghai JiaoTong University School of Medicine
Locations (1):
- Department of Hematology, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen L, Zhu HM, Li Y, Liu QF, Hu Y, Zhou JF, Jin J, Hu JD, Liu T, Wu DP, Chen JP, Lai YR, Wang JX, Li J, Li JY, Du X, Wang X, Yang MZ, Yan JS, Ouyang GF, Liu L, Hou M, Huang XJ, Yan XJ, Xu D, Li WM, Li DJ, Lou YJ, Wu ZJ, Niu T, Wang Y, Li XY, You JH, Zhao HJ, Chen Y, Shen Y, Chen QS, Chen Y, Li J, Wang BS, Zhao WL, Mi JQ, Wang KK, Hu J, Chen Z, Chen SJ, Li JM. Arsenic trioxide replacing or reducing chemotherapy in consolidation therapy for acute promyelocytic leukemia (APL2012 trial). Proc Natl Acad Sci U S A. 2021 Feb 9;118(6):e2020382118. doi: 10.1073/pnas.2020382118. PMID 33495363